CLINICAL TRIAL: NCT02552771
Title: A Randomized Trial of Mitral Valve Repair With Leaflet Resection Versus Leaflet Preservation on Functional Mitral Stenosis: The Canadian Mitral Research Alliance (CAMRA-1) Trial
Brief Title: The Canadian Mitral Research Alliance (CAMRA) Trial CardioLink-2
Acronym: CAMRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-162
Record Dates: First submitted 2015-07-30; First posted 2015-09-17 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Mitral Valve Prolapse
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mitral repair with leaflet preservation (Active Comparator): Placing man-made fibers (sutures) to more securely connect the mitral leaflets to the papillary muscles (muscles located in the ventricle).
  Interventions: Procedure: Mitral repair with leaflet preservation
- Mitral repair with leaflet resection (Active Comparator): Removal of one or both of the mitral leaflets that flop or bulge back.
  Interventions: Procedure: Mitral repair with leaflet resection

INTERVENTIONS:
Procedure: Mitral repair with leaflet preservation — Placing man-made fibers (sutures) to more securely connect the mitral leaflets to the papillary muscles (muscles located in the ventricle).
  Arms: Mitral repair with leaflet preservation
Procedure: Mitral repair with leaflet resection — Removing one or both of the mitral leaflets that flop or bulge back.
  Arms: Mitral repair with leaflet resection

SUMMARY:
Multicentre, double-armed, randomized controlled trial designed to compare mitral valve leaflet resection versus leaflet preservation with regards to the development of functional mitral stenosis following surgical repair of mitral valve prolapse. Patients will be randomized (1:1) to receive: (1) mitral valve repair with a leaflet resection or (2) mitral valve repair with leaflet preservation (using polytetrafluoroethylene neochordae), followed by echocardiographic and clinical assessment at 12-months following surgery.

DETAILED DESCRIPTION:
Mitral valve repair has emerged as the preferred surgical treatment for mitral valve prolapse (MVP), a condition wherein the mitral valve does not close properly. One common strategy for mitral valve repair is leaflet resection, which involves removing part of one or both of the mitral leaflets that flop or bulge back (prolapse). Another strategy is leaflet preservation, which involves placing man-made fibers (sutures) to more securely connect the mitral leaflets to the papillary muscles (muscles located in the ventricle). While both strategies are routinely used and lead to successful mitral valve repair, there is no clear evidence as to whether one strategy is better than the other in terms of long term outcome. The purpose of this study is to determine if one repair strategy (leaflet resection versus leaflet preservation) leads to better longer term patient outcomes. A total of 88 patients from 6 Canadian centres will be randomly assigned to one of the two strategies. The primary outcome will be functional mitral stenosis (MS) as assessed by 12-month mean mitral valve pressure gradient at peak exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with mitral regurgitation and mitral valve prolapse who are scheduled for elective mitral valve repair by an experienced mitral valve repair surgeon (>15 degenerative mitral valve repairs per year, with a repair rate>90%, and able to perform mitral repair with either a leaflet resection or leaflet preservation strategy).
2. Planned mitral valve repair amenable to either a leaflet resection or leaflet preservation surgical repair strategy

Exclusion Criteria:

1. Patients with anterior leaflet or commissural prolapse
2. Patients with endocarditis or rheumatic mitral valve disease
3. Patients with mitral annular calcification extending beyond the circumference of one leaflet scallop
4. Patients with significant LV dysfunction defined as a LVEF <40%
5. Patients undergoing concomitant aortic valve surgery
6. Patients unable to undergo bicycle ergometry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Mean mitral valve gradient at peak exercise 12-months following repair | 12 months following repair

SECONDARY OUTCOMES:
Mitral valve area | 12 months following repair
Age/Sex predicted metabolic equivalent score | 12 months following repair
Mitral leaflet coaptation height | 12 months following repair
6-minute walk test | 12 months following repair
Composite MACE (major adverse cardiovascular event) end-point of recurrent MR ≥2+, death, or hospital re-admission for congestive heart failure within 12-months of surgery | 12 months following repair

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Subodh Verma, MD, Principal Investigator — Unity Health Toronto
Locations (6):
- Canada (6):
  - Memorial University, St. John's, Newfoundland and Labrador
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec

REFERENCES:
- [Background] Theal M, Sleik K, Anand S, Yi Q, Yusuf S, Lonn E. Prevalence of mitral valve prolapse in ethnic groups. Can J Cardiol. 2004 Apr;20(5):511-5. PMID 15100753
- [Background] Freed LA, Levy D, Levine RA, Larson MG, Evans JC, Fuller DL, Lehman B, Benjamin EJ. Prevalence and clinical outcome of mitral-valve prolapse. N Engl J Med. 1999 Jul 1;341(1):1-7. doi: 10.1056/NEJM199907013410101. PMID 10387935
- [Background] Flack JM, Kvasnicka JH, Gardin JM, Gidding SS, Manolio TA, Jacobs DR Jr. Anthropometric and physiologic correlates of mitral valve prolapse in a biethnic cohort of young adults: the CARDIA study. Am Heart J. 1999 Sep;138(3 Pt 1):486-92. doi: 10.1016/s0002-8703(99)70151-1. PMID 10467199
- [Background] Ling LH, Enriquez-Sarano M, Seward JB, Tajik AJ, Schaff HV, Bailey KR, Frye RL. Clinical outcome of mitral regurgitation due to flail leaflet. N Engl J Med. 1996 Nov 7;335(19):1417-23. doi: 10.1056/NEJM199611073351902. PMID 8875918
- [Background] Enriquez-Sarano M, Avierinos JF, Messika-Zeitoun D, Detaint D, Capps M, Nkomo V, Scott C, Schaff HV, Tajik AJ. Quantitative determinants of the outcome of asymptomatic mitral regurgitation. N Engl J Med. 2005 Mar 3;352(9):875-83. doi: 10.1056/NEJMoa041451. PMID 15745978
- [Background] Verma S, Mesana TG. Mitral-valve repair for mitral-valve prolapse. N Engl J Med. 2009 Dec 3;361(23):2261-9. doi: 10.1056/NEJMct0806111. No abstract available. PMID 19955526
- [Background] Chan V, Malas T, Lapierre H, Boodhwani M, Lam BK, Rubens FD, Hendry PJ, Masters RG, Goldstein W, Mesana TG, Ruel M. Reoperation of left heart valve bioprostheses according to age at implantation. Circulation. 2011 Sep 13;124(11 Suppl):S75-80. doi: 10.1161/CIRCULATIONAHA.110.011973. PMID 21911822
- [Background] O'Brien SM, Shahian DM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 2--isolated valve surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S23-42. doi: 10.1016/j.athoracsur.2009.05.056. PMID 19559823
- [Background] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 3--valve plus coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S43-62. doi: 10.1016/j.athoracsur.2009.05.055. PMID 19559824
- [Background] Ikonomidis JS, Kratz JM, Crumbley AJ 3rd, Stroud MR, Bradley SM, Sade RM, Crawford FA Jr. Twenty-year experience with the St Jude Medical mechanical valve prosthesis. J Thorac Cardiovasc Surg. 2003 Dec;126(6):2022-31. doi: 10.1016/j.jtcvs.2003.07.005. PMID 14688722
- [Background] Chan V, Jamieson WR, Lam BK, Ruel M, Ling H, Fradet G, Mesana TG. Influence of the On-X mechanical prosthesis on intermediate-term major thromboembolism and hemorrhage: a prospective multicenter study. J Thorac Cardiovasc Surg. 2010 Nov;140(5):1053-8.e2. doi: 10.1016/j.jtcvs.2009.10.068. Epub 2010 May 23. PMID 20546795
- [Background] Chan V, Ruel M, Elmistekawy E, Mesana TG. Determinants of left ventricular dysfunction after repair of chronic asymptomatic mitral regurgitation. Ann Thorac Surg. 2015 Jan;99(1):38-42. doi: 10.1016/j.athoracsur.2014.07.025. Epub 2014 Nov 6. PMID 25442982
- [Background] Chan V, Ruel M, Hynes M, Chaudry S, Mesana TG. Impact of mitral annular calcification on early and late outcomes following mitral valve repair of myxomatous degeneration. Interact Cardiovasc Thorac Surg. 2013 Jul;17(1):120-5. doi: 10.1093/icvts/ivt163. Epub 2013 Apr 14. PMID 23587525
- [Background] Chan V, Ruel M, Chaudry S, Lambert S, Mesana TG. Clinical and echocardiographic outcomes after repair of mitral valve bileaflet prolapse due to myxomatous disease. J Thorac Cardiovasc Surg. 2012 Apr;143(4 Suppl):S8-11. doi: 10.1016/j.jtcvs.2012.01.046. Epub 2012 Feb 4. PMID 22306213
- [Background] Castillo JG, Anyanwu AC, Fuster V, Adams DH. A near 100% repair rate for mitral valve prolapse is achievable in a reference center: implications for future guidelines. J Thorac Cardiovasc Surg. 2012 Aug;144(2):308-12. doi: 10.1016/j.jtcvs.2011.12.054. Epub 2012 Jun 12. PMID 22698565
- [Background] Carpentier A. Cardiac valve surgery--the "French correction". J Thorac Cardiovasc Surg. 1983 Sep;86(3):323-37. No abstract available. PMID 6887954
- [Background] Braunberger E, Deloche A, Berrebi A, Abdallah F, Celestin JA, Meimoun P, Chatellier G, Chauvaud S, Fabiani JN, Carpentier A. Very long-term results (more than 20 years) of valve repair with carpentier's techniques in nonrheumatic mitral valve insufficiency. Circulation. 2001 Sep 18;104(12 Suppl 1):I8-11. PMID 11568021
- [Background] Filsoufi F, Carpentier A. Principles of reconstructive surgery in degenerative mitral valve disease. Semin Thorac Cardiovasc Surg. 2007 Summer;19(2):103-10. doi: 10.1053/j.semtcvs.2007.04.003. PMID 17870003
- [Background] Kuperstein R, Spiegelstein D, Rotem G, Stein M, Kogan A, Sternik L, Raanani E. Late clinical outcome of transient intraoperative systolic anterior motion post mitral valve repair. J Thorac Cardiovasc Surg. 2015 Feb;149(2):471-6. doi: 10.1016/j.jtcvs.2014.10.043. Epub 2014 Oct 14. PMID 25454906
- [Background] Seeburger J, Falk V, Borger MA, Passage J, Walther T, Doll N, Mohr FW. Chordae replacement versus resection for repair of isolated posterior mitral leaflet prolapse: a egalite. Ann Thorac Surg. 2009 Jun;87(6):1715-20. doi: 10.1016/j.athoracsur.2009.03.003. PMID 19463584
- [Background] Falk V, Seeburger J, Czesla M, Borger MA, Willige J, Kuntze T, Doll N, Borger F, Perrier P, Mohr FW. How does the use of polytetrafluoroethylene neochordae for posterior mitral valve prolapse (loop technique) compare with leaflet resection? A prospective randomized trial. J Thorac Cardiovasc Surg. 2008 Nov;136(5):1205; discussion 1205-6. doi: 10.1016/j.jtcvs.2008.07.028. Epub 2008 Sep 14. PMID 19026803
- [Background] Lange R, Guenther T, Noebauer C, Kiefer B, Eichinger W, Voss B, Bauernschmitt R, Tassani-Prell P, Mazzitelli D. Chordal replacement versus quadrangular resection for repair of isolated posterior mitral leaflet prolapse. Ann Thorac Surg. 2010 Apr;89(4):1163-70; discussion 1170. doi: 10.1016/j.athoracsur.2009.12.057. PMID 20338326
- [Background] Nishimura RA, Otto CM, Bonow RO, Carabello BA, Erwin JP 3rd, Guyton RA, O'Gara PT, Ruiz CE, Skubas NJ, Sorajja P, Sundt TM 3rd, Thomas JD; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC guideline for the management of patients with valvular heart disease: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 10;63(22):2438-88. doi: 10.1016/j.jacc.2014.02.537. Epub 2014 Mar 3. No abstract available. PMID 24603192
- [Background] Chan KL, Chen SY, Chan V, Hay K, Mesana T, Lam BK. Functional significance of elevated mitral gradients after repair for degenerative mitral regurgitation. Circ Cardiovasc Imaging. 2013 Nov;6(6):1041-7. doi: 10.1161/CIRCIMAGING.112.000688. Epub 2013 Sep 6. PMID 24014825
- [Background] Mesana TG, Lam BK, Chan V, Chen K, Ruel M, Chan K. Clinical evaluation of functional mitral stenosis after mitral valve repair for degenerative disease: potential affect on surgical strategy. J Thorac Cardiovasc Surg. 2013 Dec;146(6):1418-23; discussion 1423-5. doi: 10.1016/j.jtcvs.2013.08.011. Epub 2013 Sep 26. PMID 24075470
- [Background] Gammie JS, Sheng S, Griffith BP, Peterson ED, Rankin JS, O'Brien SM, Brown JM. Trends in mitral valve surgery in the United States: results from the Society of Thoracic Surgeons Adult Cardiac Surgery Database. Ann Thorac Surg. 2009 May;87(5):1431-7; discussion 1437-9. doi: 10.1016/j.athoracsur.2009.01.064. PMID 19379881
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Derived] Rumman RK, Verma S, Chan V, Fottinger A, Quan A, Hibino M, de Varennes BE, Burns DJP, Chu MWA, Teoh H, Latter DA, Bisleri G, Leong-Poi H, Mazer CD, Connelly KA. Comparison of myocardial mechanics after mitral valve repair with leaflet preservation versus leaflet resection: A subanalysis of the randomized Canadian Mitral Research Alliance CardioLink-2 trial. J Thorac Cardiovasc Surg. 2025 Aug 7:S0022-5223(25)00654-3. doi: 10.1016/j.jtcvs.2025.07.047. Online ahead of print. PMID 40783073
- [Derived] Rumman RK, Verma S, Chan V, Mazer D, Quan A, Hibino M, De Varennes B, Chu MWA, Latter D, Teoh H, Yanagawa B, Leong-Poi H, Connelly KA. Predictors of mitral valve haemodynamics after mitral valve repair for degenerative mitral regurgitation. Heart. 2023 May 15;109(11):866-873. doi: 10.1136/heartjnl-2022-321753. PMID 36750353
- [Derived] Chan V, Mazer CD, Ali FM, Quan A, Ruel M, de Varennes BE, Gregory AJ, Bouchard D, Whitlock RP, Chu MWA, Dokollari A, Mesana T, Bhatt DL, Latter DA, Zuo F, Tsang W, Teoh H, Juni P, Leong-Poi H, Verma S. Randomized, Controlled Trial Comparing Mitral Valve Repair With Leaflet Resection Versus Leaflet Preservation on Functional Mitral Stenosis: The CAMRA CardioLink-2 Study. Circulation. 2020 Oct 6;142(14):1342-1350. doi: 10.1161/CIRCULATIONAHA.120.046853. Epub 2020 Oct 5. PMID 33017212
- [Derived] Chan V, Chu MWA, Leong-Poi H, Latter DA, Hall J, Thorpe KE, de Varennes BE, Quan A, Tsang W, Dhingra N, Yared K, Teoh H, Chu FV, Chan KL, Mesana TG, Connelly KA, Ruel M, Juni P, Mazer CD, Verma S. Randomised trial of mitral valve repair with leaflet resection versus leaflet preservation on functional mitral stenosis (The CAMRA CardioLink-2 Trial). BMJ Open. 2017 May 30;7(5):e015032. doi: 10.1136/bmjopen-2016-015032. PMID 28566364